CLINICAL TRIAL: NCT05979714
Title: Developing a Novel Delivery System for CAB-RPV LA in Transgender Women Living With HIV in Public Health Settings
Brief Title: The Cheeky Study: A Novel Delivery System for CAB-RPV LA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: ViiV Healthcare (Industry); San Francisco Department of Public Health (Other Government); Lyon-Martin Community Health Services (Unknown)
Responsible Party: Principal Investigator, Albert Liu, Clinical Research Director, Public Health Foundation Enterprises, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-35957
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections
Keywords: Transwomen
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: This study proposes using mixed methods to tailor and evaluate implementation and client outcomes when CAB-RPV LA is delivered through this integrated delivery model. Our approach will be guided by a rigorous implementation science approach using the Proctor Model to evaluate our implementation strategies.
  The Proctor Model posits that improvements in outcomes are dependent on the evidence-based intervention selected for implementation and on the strategies used to deliver the intervention. The model distinguishes between the intervention (CAB-RPV LA), different types of implementation strategies, and different levels of outcomes that are expected to build on each other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cheeky Study Intervention (Experimental): This study represents a hybrid design type 3 focusing primarily on implementation outcomes and secondarily on clinical effectiveness among trans women living with HIV receiving care within primary care clinics in San Francisco. A type 3 design was chosen, as the clinical efficacy of CAB- RPV LA has been established in clinical trials, and the focus of this study is on initial implementation of CAB-RPV LA within these clinics.
  Interventions: Other: Patient-centered injection site; Behavioral: Patient-centered adherence support; Other: Provider education; Behavioral: Improved clinic communication strategies

INTERVENTIONS:
Other: Patient-centered injection site — CAB-RPV LA will be delivered in a trans-friendly injection clinic at Bridge HIV, which is centrally located in SF. The clinic is staffed by physicians, nurses, and peer navigators who are experienced working with the trans community and are experts in delivery of injectable formulations. For patients unable to attend follow-up clinic visits, arrangements will be made for a clinical provider and peer navigator to conduct a home visit for injection delivery. This implementation strategy will overcome structural barriers where it is difficult to get a visit appointment, and when appointments are missed, even harder to re-schedule. The central location in a quiet, safe and trans-affirming clinical site will make injections easy-to-access. Because the Bridge HIV clinic is not a primary care site, injections can be delivered with minimal wait times due to low patient load relative to clinical capacity.
Behavioral: Patient-centered adherence support — A Trans peer navigator will support trans women living with HIV receiving long-acting injectable treatment through our delivery model. Peer navigators will reach out to trans women using our highly effective mobile SMS platform to provide additional support before and between visits. This platform provides automated weekly check-ins for streamlined support and bi-directional asynchronous texting with a peer navigator. Peer navigators will use this SMS platform to send appointment reminders, assess needs for re-scheduling, answer questions and triage concerns regarding CAB-RPV LA, and offer support for transportation or scheduling a home visit. This approach has demonstrated efficacy in improving ART adherence and viral suppression in people living with HIV as well as retention in care and adherence to PrEP.
Other: Provider education — To support effective outreach to and education of providers on novel evidence-based practices, SFDPH has utilized public health detailing (brief educational visits via a nurse practitioner) to ensure providers are prepared to implement new interventions. This strategy has been effective in expanding the implementation of PrEP, RAPID ART initiation, and comprehensive STI screening across clinics in SF. For this study, we will develop educational materials on the CAB-RPV LA regimen, including a summary of results from Phase 3 trials (ATLAS20, FLAIR21), the FDA labeling indication, and details about SFDPH's implementation of CAB-RPV LA within our safety-net system and our new delivery model. These materials will include information on which patients will be eligible for this treatment modality and eligible for referral to our new delivery model, and how to make these referrals.
Behavioral: Improved clinic communication strategies — For SFDPH clinics, Bridge HIV providers will communicate with primary care providers through EPIC, SFDPH's electronic health record (EHR), and one of the most common EHR systems used across clinic systems in the US. For this study, secure email and/or telephone encounters within EPIC will be used to facilitate efficient referrals of TGW living with HIV from their primary providers to the Bridge HIV injection clinic and ongoing secure communication between Bridge HIV clinicians and the primary care team. For non-SFDPH clinics, communication will be via secure email or other secure communication strategies.

SUMMARY:
This is a single-arm implementation study of a novel integrated delivery model of CAB-RPV LA for transwomen living with HIV.

DETAILED DESCRIPTION:
CAB-RPV LA as a monthly injectable could address disparities in viral suppression among trans women living with HIV. This study is designed to enroll a diverse population of trans women living with HIV who receive HIV care within collaborating primary care clinics. This study proposes using mixed methods to tailor and evaluate implementation and client outcomes when CAB-RPV LA is delivered through this integrated delivery model.

This will be a 9-month pilot study among 40 participants who will be provided CAB-RPV LA through an integrated trans-friendly delivery model using 4 implementation strategies to improve the adoption and integration of CAB-RPV LA delivery to trans women. These strategies are aimed at all levels of implementation - system, clinic, provider, and patient to maximize impact. The 4 strategies are a patient-centered injection site (Bridge HIV, SFDPH), patient-centered adherence support (peer health navigation and SMS platform with reminders and communication with staff), provider education, and improved clinic communication strategies.. CAB-RPV LA is being provided as standard of care and is not paid for by the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Male sex at birth and gender identity other than male
* Willing and able to provide written informed consent
* HIV-infected, confirmed by laboratory testing (can be via medical record)
* Eligible to receive CAB-RPV LA per FDA-approved label
* Virologically suppressed at the last visit within the last 6 months (HIV RNA <50 copies/ml)
* Interested in initiating CAB-RPV LA for HIV treatment and willing to receive injections at Bridge HIV
* Currently receiving HIV care by a care provider at one of the collaborating primary care clinics.
* Has a cell phone and active service
* Able to understand, read, and speak English

Exclusion Criteria:

* Unable to receive gluteal injections
* Plans to move away from the site area within the next 9 months.
* History of known or suspected drug resistance that would compromise the CAB-RPV regimen

  * Rilpivirine: L100I; K101E; V106I and A; V108I; E138K and A, G, Q, R; V179F and I; Y181C and I; V189I; G190E; H221Y and H/L; F227C; and M230I and L; K103N+K238T, K103N+E138G+K238T; Y188L
  * Cabotegravir: Q146L; S153Y; I162M; T124A; Q148H, K; C56S; V72I; L74M; V75A; T122N; E138K; G140S; G149A; M154I; and N155H
* Prior hypersensitivity to cabotegravir or rilpivirine
* Current or expected use of any of the following medications:

  * Anticonvulsants: carbamazepine, oxcarbazepine, phenobarbital, phenytoin
  * Antimycobacterials: rifabutin, rifampin, rifapentine
  * Systemic glucocorticoids: more than a single dose of dexamethasone
  * Herbal: St John's Wort
* Any medical, psychiatric, or social condition or other responsibilities that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — transgender women
Enrollment: 50 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of delivering CAB-RPV LA | 0, 9,18 Months
  Assess the feasibility of delivering CAB-RPV LA to trans women living with HIV via a trans-tailored, integrated delivery model
Acceptability of delivering CAB-RPV LA | 0, 9,18 Months
  Assess the acceptability of delivering CAB-RPV LA to trans women living with HIV via a trans-tailored, integrated delivery model
Client Satisfaction | 0, 3, 6, 9 Months
  Assess client satisfaction with treatment when CAB-RPV LA is delivered through a trans-tailored integrated model

SECONDARY OUTCOMES:
Assess tolerability | 3, 6, 9 Months
  Assess tolerability of CAB-RPV LA among trans women receiving CAB-LA injections
Assess adherence to injections | 3, 6, 9 Months
  Assess adherence to monthly or bimonthly injections among trans women receiving CAB-RPV LA in this delivery model
Assess viral suppression | 3, 6, 9 Months
  Assess viral suppression rates among trans women receiving CAB-RPV LA
Describe development of resistance mutations | 3, 6, 9 Months
  Describe development of resistance mutations in cases of virologic failure among trans women receiving CAB-RPV LA

CONTACTS AND LOCATIONS:
Overall Officials: Albert Liu, MD, MPH, Principal Investigator — SFDPH Bridge HIV
Locations (1):
- Bridge HIV, San Francisco Department of Public Health, San Francisco, California, United States